CLINICAL TRIAL: NCT00006255
Title: A Phase II Study of Magnetic Resonance Guided and Monitored Interstitial Thermal Radiofrequency Ablation of Primary Renal Cell Carcinoma, Hepatic Metastasis, and Other Sites of Solid Organ Tumor and Metastases
Brief Title: Magnetic Resonance Imaging-guided Thermal Radiofrequencey Ablation of Primary Renal Cell Carcinoma, Hepatic Metastasis, and Other Sites of Solid Organ Tumor and Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John R. Haaga, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2Y00; P30CA043703 (NIH); CWRU-2Y00; NCI-G00-1850
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Kidney Cancer; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; unspecified adult solid tumor, protocol specific; liver metastases
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radiofrequency ablation — Undergo thermal ablation by radiofrequency energy under magnetic resonance guidance.Thermal ablation continues until the entire tumor is treated.
Procedure: thermal ablation therapy — Undergo thermal ablation by radiofrequency energy under magnetic resonance guidance.Thermal ablation continues until the entire tumor is treated.

SUMMARY:
RATIONALE: Radiofrequency ablation uses high-frequency electric current to heat and kill tumor cells. Magnetic resonance imaging-guided radiofrequency ablation may an effective treatment for primary kidney cancer, liver metastases, or other solid tumors.

PURPOSE: Phase II trial to study the effectiveness of magnetic-resonance-guided radiofrequency ablation in treating patients who have primary kidney cancer, liver metastases, or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether magnetic resonance image monitoring during radiofrequency interstitial thermal ablation can accurately predict complete destruction of focal tumor along with an adequate margin of normal tissue, as demonstrated by absence of growth on subsequent imaging studies for a 1-year period, in patients with primary renal cell carcinoma, hepatic metastases, or other solid tumors.

OUTLINE: Patients are stratified according to disease (localized hepatic metastases vs primary renal neoplasms vs solid tumors in other sites).

Patients undergo thermal ablation by radiofrequency energy under magnetic resonance guidance. Thermal ablation continues until the entire tumor is treated. Treatment ceases when the entire lesion has undergone necrosis or the zone of necrosis or significant heat deposition approaches vital neurovascular structures.

Patients are followed at 2 weeks and at 3, 6, 9, and 12 months.

PROJECTED ACCRUAL: A total of 28-39 patients will be accrued for this study within 22-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary renal cell carcinoma, hepatic metastases, or other solid tumor meeting the following criteria:

  * Not amenable to curative or substantial palliative therapy OR
  * Failed chemotherapy or biological response modifier therapy OR
  * Unlikely to benefit from conventional chemotherapy
  * No more than 5 measurable metastatic masses in the liver

    * No greater than 5 cm in diameter
  * Other tumor sites allowed if location and size amenable to ablation therapy
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 4 months

Hematopoietic:

* Granulocyte count at least 1,000/mm^3
* Hemoglobin at least 8.0 g/dL
* Platelet count at least 100,000/mm^3
* No untreated bleeding diathesis

Hepatic:

* PT no greater than 13.5 seconds
* PT/PTT normal if prior warfarin or heparin use

Renal:

* Not specified

Cardiovascular:

* No implanted pacemaker, incompatible aneurysm clip, or other device that would preclude magnetic resonance imaging
* No myocardial infarction within the past 6 weeks
* No unstable angina

Other:

* Not pregnant or nursing
* No serious active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 28 days since prior biological response modifier therapy

Chemotherapy:

* See Disease Characteristics
* At least 28 days since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to study lesion

Surgery:

* Not specified

Other:

* At least 7 days since prior nonsteroidal antiinflammatory drugs or aspirin
* At least 1 hour since prior heparin
* No concurrent warfarin
* No concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2000-04; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Determine whether magnetic resonance image monitoring during radiofrequency interstitial thermal ablation can accurately predict complete destruction of focal tumor along with an adequate margin of normal tissue. | Patients are followed at 2 weeks and at 3, 6, 9, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: John R. Haaga, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States